CLINICAL TRIAL: NCT03629548
Title: Comparing Combined Foley Catheter Balloon and PGE2 Vaginal Ovule With Early Amniotomy and PGE2 for Induction of Labor at Term: A Randomized Study
Brief Title: Comparing Foley Catheter Balloon With Early Amniotomy for Induction of Labor at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, Principal investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48
Record Dates: First submitted 2018-03-27; First posted 2018-08-14 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Induced Vaginal Delivery
Keywords: dinoprostone; early amniotomy; labor induction; foley bulb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early amniotomy plus dinoprostone (Active Comparator): 10 mg dinoprostone vaginal ovul will be inserted to the posterior fornix. Early amniotomy will be done in the early active phase of labor for early amniotomy group ( half of participants) when the cervix will be dilated 3 cm using the amniotomy hook.
  Interventions: Procedure: early amniotomy
- foley balloon catheter plus dinoprostone (Experimental): an 18-F Foley catheter which filling with 30 mL of saline solution will be placed into the cervix and after placement of balloon catheter 10 mg dinoprostone vaginal ovul will be inserted to the posterior fornix
  Interventions: Device: foley catheter balloon placement

INTERVENTIONS:
Procedure: early amniotomy — 10 mg PGE2 vaginal ovul will be inserted to the posterior fornix. Early amniotomy will be done in the early active phase of labor for early amniotomy group ( half of participants) when the cervix will be dilated 3 cm using the amniotomy hook.
  Arms: early amniotomy plus dinoprostone
Device: foley catheter balloon placement — an 18-F Foley catheter which filling with 30 mL of saline solution will be placed into the cervix and after placement of balloon catheter 10 mg PGE2 vaginal ovul will be inserted to the posterior fornix
  Other Names: mechanic and medical method
  Arms: foley balloon catheter plus dinoprostone

SUMMARY:
This study evaluates the intervention for induction of labor with low bishop scores . One group will be induced by transcervical Foley catheter balloon and vaginal PGE2 and other group will be induced by early amniotomy and PGE2 vaginal ovule for induction of labor at term.

DETAILED DESCRIPTION:
An unfavorable cervix during induction decreases the success rate of labor induction and vaginal delivery. Therefore it is required to apply cervical ripening methods for unfavorable cervices. Application of transcervical Foley catheter is an effective mechanical method and has the advantages of lower cost and lowest rate of fetal heart rate changes due to tachysystole compared with PGE1 and PGE2. Despite the advantages of mechanical methods, PGE1 and PGE2 are reported to be more effective than mechanical methods to achieve vaginal delivery within 24 hours. Although there are a lot of studies comparing PGE1, PGE2 and transcervical Foley balloon catheter separately and PGE1 combined with transcervical Foley balloon catheter, less is known about combined usage of PGE2 and transcervical Foley balloon catheter. Early amniotomy is another effective method to ripen cervix. we aim to evaluate which method is superior to another.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy,
2. gestational age ≥37 weeks,
3. intact membranes,
4. cephalic presentation,
5. bishop score ≤5,
6. had obstetrical indications for induction of labor,
7. had less than three uterine contractions in every 10 minutes.

Exclusion Criteria:

1. Patients who had contraindications for vaginal delivery,
2. previous uterine surgery,
3. fetal malpresentation,
4. multifetal pregnancy,
5. more than three contractions in 10 minutes,
6. contraindications to prostaglandins,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — term pregnancies
Enrollment: 250 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
induction-to- delivery time | from the beginning of induction until the labor
  the length of time between the beginning of induction and the end of labor

SECONDARY OUTCOMES:
induction-to-active phase of labor time | from the beginning of induction until the labor
  the length of time between the beginning of induction and the onset of labor

CONTACTS AND LOCATIONS:
Overall Officials: ahmet eser, M.D., Study Director — Zeynep Kamil Maternity and Children's Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey
Locations (1):
- Zeynep Kamil Education and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264